CLINICAL TRIAL: NCT04787731
Title: Efficacy of Two Dental Local Anesthetics on the Oral Health-Related Quality of Life After Endodontic Treatment in the Symptomatic Mandibular Molars: A Double Blind Randomized Controlled Trial
Brief Title: Efficacy of Two Local Anesthetics on Quality of Life After Endodontic Treatment
Acronym: B-OHIP14
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: COVID-19 and Personnel changes
Sponsor: NYU College of Dentistry (Other)
Responsible Party: Principal Investigator, Asgeir Sigurdsson, DDS, MS, Professor and Chair Department of Endodontics, NYU College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: s19-00069
Record Dates: First submitted 2021-03-04; First posted 2021-03-09 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Pain, Postoperative; Quality of Life
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Double blind randomized clinical trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocaine HCI (1.7mL) 2% concentration with epinephrine (1:100,000) is the control agent. It exists in liquid form in cartridges. Lidocaine is a FDA approved marketed anesthetic drug.
  Interventions: Drug: Bupivacaine Local Anesthetic
- Bupivacaine (Active Comparator): Bupivacaine HCI (1.8mL) 5% concentration, with epinephrine (1:200,000) is the investigational product. It exists in liquid form in cartridges. Bupivacaine is a FDA approved marketed anesthetic drug and meets IND Exemption.
  Interventions: Drug: Bupivacaine Local Anesthetic

INTERVENTIONS:
Drug: Bupivacaine Local Anesthetic — Long lasting local anesthetic administered to be compared to Lidocaine for quality of life outcomes in dental patients undergoing endodontic treatment
  Other Names: Lidocaine Local Anesthetic

SUMMARY:
In this randomized controlled double-blinded study, subjects will be assigned to one of two study groups to either be anesthetized with Bupivacaine or Lidocaine prior to needed treatment of pulpectomy/endodontic debridement on a symptomatic tooth.

Subjects' oral health related quality of life and postoperative pain resolution, pain medication use and numbness will be compared in two study groups.

DETAILED DESCRIPTION:
This is a double-blind randomized controlled single-site trial. We aim to recruit 100 subject, with an anticipated dropout rate of 20%; our goal is to enroll 40 subjects in each study arm based on the power analysis described in data analysis section as well as general feasibility for recruitment, and the ability to complete the study in within one year.

After screening for eligibility based on the inclusion and exclusion criteria listed below, and after preoperative data collection, in the experimental arm, inferior alveolar nerve block (IANB) will be administered 0.5% bupivacaine with 1:200,000 epinephrine whereas in the control arm, IANB will be administered 2% lidocaine with 1:100,000 epinephrine for a standardized pulpectomy/endodontic debridement treatment as the 1st visit endodontic treatment for subjects with preoperative pain. Postoperative oral health related quality of life questionnaire (OHIP-14) responses at day 1 and 5 as well as 5-day postoperative pain intensity questionnaire will be collected remotely. In this way, we will be able to compare OHQoL change as well as postoperative pain resolution, pain medication use and postoperative soft tissue anesthesia reported by the patient in two study arms.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18-85 years
* Patients with pulpal diagnosis of either symptomatic irreversible pulpitis or pulp necrosis and periapical diagnosis of normal apical tissues, symptomatic apical periodontitis or asymptomatic apical periodontitis.
* Patients who only have one tooth with odontogenic pain at the time point of the screening.
* Patients who are treatment planned, and have agreed to have, pulpectomy/endodontic debridement.
* Patients with acute dental pain of at least 3/10 on NRS
* Patients must be able to comprehend and complete all study questionnaires
* Patients must be able to comprehend the description of the study protocol and written consent Patients must be able to be contacted by text messages, phone calls or email during 5 days after pulpectomy/endodontic debridement

Exclusion Criteria:

* Medically complex patients with severe systemic diseases (ASA III or above). These may include uncontrolled diabetes, uncontrolled blood pressure and/or chronic renal failure, for example, and potential participants will be asked about these conditions during the screening process.
* Pregnant Patients
* Patients who have already been enrolled in the study. Patients can only be enrolled for treatment on one tooth.
* Patients with known hypersensitivity or allergy to any local anesthetic agent of the amide group, or any other components of the two anesthetic solutions such as epinephrine, sodium metabisulfite used in the study.
* Patients who use ergot-type oxytocic drugs for uterine contraction, monoamine oxidase inhibitors, antidepressant of triptyline or imipramine types or patients who are planned to receive sedatives for the treatment.
* Patients with additional elective dental treatments like extraction, implant placement, root canal therapy planned in the 5 days following the date of enrollment in this study
* Patients with pain whose examined tooth is planned for vital pulp therapies e.g. pulpotomy, retreatment, apical surgery or extraction
* Patients with a pulpal diagnosis or reversible pulpitis, previously treated, previously initiated therapy and periapical diagnosis of acute apical abscess or chronic apical abscess.
* Patients who have multiple teeth with odontogenic pain at the time of the screening
* Patients who do not understand or are able to read the questionnaires
* Non-English speaking patients

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Effects of Bupivacaine/Lidocaine will be assessed on post-operative pain intensity, medication use and length of numbness compared between the two study groups using Oral Health Related Quality-of-Life (OHQoL) questionnaire and Visual Analog Scale (VAS). | 4 weeks +-10 days
  The OHQoL questionnaire contains 14 questions and scores can range from 0 to 56. Pain intensity is measured by VAS scale and scores can range from 0-10. Higher scores represent worse outcomes for both assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Asgeir Sigurdsson, Principal Investigator — NYU Dentistry
Locations (1):
- NYU College of Dentistry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pak JG, White SN. Pain prevalence and severity before, during, and after root canal treatment: a systematic review. J Endod. 2011 Apr;37(4):429-38. doi: 10.1016/j.joen.2010.12.016. PMID 21419285
- [Background] Arias A, de la Macorra JC, Hidalgo JJ, Azabal M. Predictive models of pain following root canal treatment: a prospective clinical study. Int Endod J. 2013 Aug;46(8):784-93. doi: 10.1111/iej.12059. Epub 2013 Feb 12. PMID 23402273
- [Background] Law AS, Nixdorf DR, Aguirre AM, Reams GJ, Tortomasi AJ, Manne BD, Harris DR; National Dental PBRN Collaborative Group. Predicting severe pain after root canal therapy in the National Dental PBRN. J Dent Res. 2015 Mar;94(3 Suppl):37S-43S. doi: 10.1177/0022034514555144. Epub 2014 Oct 29. PMID 25355775
- [Background] Rechenberg DK, Held U, Burgstaller JM, Bosch G, Attin T. Pain levels and typical symptoms of acute endodontic infections: a prospective, observational study. BMC Oral Health. 2016 May 27;16(1):61. doi: 10.1186/s12903-016-0222-z. PMID 27234432
- [Background] Owatz CB, Khan AA, Schindler WG, Schwartz SA, Keiser K, Hargreaves KM. The incidence of mechanical allodynia in patients with irreversible pulpitis. J Endod. 2007 May;33(5):552-6. doi: 10.1016/j.joen.2007.01.023. Epub 2007 Mar 6. PMID 17437870
- [Background] Khan AA, Owatz CB, Schindler WG, Schwartz SA, Keiser K, Hargreaves KM. Measurement of mechanical allodynia and local anesthetic efficacy in patients with irreversible pulpitis and acute periradicular periodontitis. J Endod. 2007 Jul;33(7):796-9. doi: 10.1016/j.joen.2007.01.021. Epub 2007 Mar 26. PMID 17804314
- [Background] Menhinick KA, Gutmann JL, Regan JD, Taylor SE, Buschang PH. The efficacy of pain control following nonsurgical root canal treatment using ibuprofen or a combination of ibuprofen and acetaminophen in a randomized, double-blind, placebo-controlled study. Int Endod J. 2004 Aug;37(8):531-41. doi: 10.1111/j.1365-2591.2004.00836.x. PMID 15230906
- [Background] Joseph P. Crowley CoADA. ADA wants Federal agencies to address Best Practices for managing acute pain. In: Vanilla M. Singh PMBPI-ATF, editor.: American Dental; Association; 2018.
- [Background] Shamszadeh S, Shirvani A, Eghbal MJ, Asgary S. Efficacy of Corticosteroids on Postoperative Endodontic Pain: A Systematic Review and Meta-analysis. J Endod. 2018 Jul;44(7):1057-1065. doi: 10.1016/j.joen.2018.03.010. Epub 2018 Apr 30. PMID 29709296
- [Background] Su N, Wang H, Zhang S, Liao S, Yang S, Huang Y. Efficacy and safety of bupivacaine versus lidocaine in dental treatments: a meta-analysis of randomised controlled trials. Int Dent J. 2014 Feb;64(1):34-45. doi: 10.1111/idj.12060. Epub 2013 Oct 11. PMID 24117122
- [Background] Parirokh M, Yosefi MH, Nakhaee N, Manochehrifar H, Abbott PV, Reza Forghani F. Effect of bupivacaine on postoperative pain for inferior alveolar nerve block anesthesia after single-visit root canal treatment in teeth with irreversible pulpitis. J Endod. 2012 Aug;38(8):1035-9. doi: 10.1016/j.joen.2012.04.012. Epub 2012 May 30. PMID 22794202
- [Background] Moradi S, Naghavi N. Comparison of bupivacaine and lidocaine use for postoperative pain control in endodontics. Iran Endod J. 2010 Winter;5(1):31-5. Epub 2010 Feb 20. PMID 24778680
- [Background] Gordon SM, Mischenko AV, Dionne RA. Long-acting local anesthetics and perioperative pain management. Dent Clin North Am. 2010 Oct;54(4):611-20. doi: 10.1016/j.cden.2010.06.002. PMID 20831925
- [Background] Balocco AL, Van Zundert PGE, Gan SS, Gan TJ, Hadzic A. Extended release bupivacaine formulations for postoperative analgesia: an update. Curr Opin Anaesthesiol. 2018 Oct;31(5):636-642. doi: 10.1097/ACO.0000000000000648. PMID 30074492
- [Background] Sampaio RM, Carnaval TG, Lanfredi CB, Horliana AC, Rocha RG, Tortamano IP. Comparison of the anesthetic efficacy between bupivacaine and lidocaine in patients with irreversible pulpitis of mandibular molar. J Endod. 2012 May;38(5):594-7. doi: 10.1016/j.joen.2012.01.008. Epub 2012 Feb 4. PMID 22515885
- [Background] Fernandez C, Reader A, Beck M, Nusstein J. A prospective, randomized, double-blind comparison of bupivacaine and lidocaine for inferior alveolar nerve blocks. J Endod. 2005 Jul;31(7):499-503. doi: 10.1097/01.don.0000167395.61075.38. PMID 15980707
- [Background] Aggarwal V, Singla M, Miglani S. Comparative Evaluation of Anesthetic Efficacy of 2% Lidocaine, 4% Articaine, and 0.5% Bupivacaine on Inferior Alveolar Nerve Block in Patients with Symptomatic Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial. J Oral Facial Pain Headache. 2017 Spring;31(2):124-128. doi: 10.11607/ofph.1642. PMID 28437508
- [Background] Parirokh M, Yosefi MH, Nakhaee N, Abbott PV, Manochehrifar H. The success rate of bupivacaine and lidocaine as anesthetic agents in inferior alveolar nerve block in teeth with irreversible pulpitis without spontaneous pain. Restor Dent Endod. 2015 May;40(2):155-60. doi: 10.5395/rde.2015.40.2.155. Epub 2015 Mar 16. PMID 25984478
- [Background] St George G, Morgan A, Meechan J, Moles DR, Needleman I, Ng YL, Petrie A. Injectable local anaesthetic agents for dental anaesthesia. Cochrane Database Syst Rev. 2018 Jul 10;7(7):CD006487. doi: 10.1002/14651858.CD006487.pub2. PMID 29990391
- [Background] Montero J, Lorenzo B, Barrios R, Albaladejo A, Miron Canelo JA, Lopez-Valverde A. Patient-centered Outcomes of Root Canal Treatment: A Cohort Follow-up Study. J Endod. 2015 Sep;41(9):1456-61. doi: 10.1016/j.joen.2015.06.003. Epub 2015 Jul 26. PMID 26211565
- [Background] Hamasha AA, Hatiwsh A. Quality of life and satisfaction of patients after nonsurgical primary root canal treatment provided by undergraduate students, graduate students and endodontic specialists. Int Endod J. 2013 Dec;46(12):1131-9. doi: 10.1111/iej.12106. Epub 2013 Apr 6. PMID 23560436
- [Background] Slade GD. Derivation and validation of a short-form oral health impact profile. Community Dent Oral Epidemiol. 1997 Aug;25(4):284-90. doi: 10.1111/j.1600-0528.1997.tb00941.x. PMID 9332805
- [Background] Chou R, Gordon DB, de Leon-Casasola OA, Rosenberg JM, Bickler S, Brennan T, Carter T, Cassidy CL, Chittenden EH, Degenhardt E, Griffith S, Manworren R, McCarberg B, Montgomery R, Murphy J, Perkal MF, Suresh S, Sluka K, Strassels S, Thirlby R, Viscusi E, Walco GA, Warner L, Weisman SJ, Wu CL. Management of Postoperative Pain: A Clinical Practice Guideline From the American Pain Society, the American Society of Regional Anesthesia and Pain Medicine, and the American Society of Anesthesiologists' Committee on Regional Anesthesia, Executive Committee, and Administrative Council. J Pain. 2016 Feb;17(2):131-57. doi: 10.1016/j.jpain.2015.12.008. PMID 26827847
- [Background] Shahi S, Rahimi S, Yavari HR, Ghasemi N, Ahmadi F. Success Rate of 3 Injection Methods with Articaine for Mandibular First Molars with Symptomatic Irreversible Pulpitis: A CONSORT Randomized Double-blind Clinical Trial. J Endod. 2018 Oct;44(10):1462-1466. doi: 10.1016/j.joen.2018.07.010. Epub 2018 Aug 31. PMID 30174101
- [Background] Shapiro MR, McDonald NJ, Gardner RJ, Peters MC, Botero TM. Efficacy of Articaine versus Lidocaine in Supplemental Infiltration for Mandibular First versus Second Molars with Irreversible Pulpitis: A Prospective, Randomized, Double-blind Clinical Trial. J Endod. 2018 Apr;44(4):523-528. doi: 10.1016/j.joen.2017.10.003. Epub 2018 Feb 1. PMID 29397214
- [Background] Hargreaves KM, Berman L. H. Cohen's Pathways of the Pulp. Missouri:Elsevier;2016
- [Background] Olmedo-Gaya MV, Manzano-Moreno FJ, Munoz-Lopez JL, Vallecillo-Capilla MF, Reyes-Botella C. Double-blind, randomized controlled clinical trial on analgesic efficacy of local anesthetics articaine and bupivacaine after impacted third molar extraction. Clin Oral Investig. 2018 Dec;22(9):2981-2988. doi: 10.1007/s00784-018-2386-1. Epub 2018 Feb 15. PMID 29450738

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT04787731/Prot_SAP_000.pdf